CLINICAL TRIAL: NCT01313325
Title: Hippotherapy to Improve Balance Deficits in a Cohort of Children With Movement Disorders: A Pilot Study
Brief Title: Hippotherapy to Improve the Balance of Children With Movement Disorders
Acronym: HPOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Central Michigan University (Other)
Responsible Party: Dr. Debbie Silkwood-Sherer, Central Michigan University
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 09/14/2006
Record Dates: First submitted 2011-03-09; First posted 2011-03-11 (Estimated); Last update posted 2011-03-11 (Estimated); Status verified 2011-03

CONDITIONS: Neuromuscular Diseases; Cerebral Palsy; Down Syndrome; Autism; Developmental Coordination Disorder
Keywords: hippotherapy; neuromuscular disorders; balance deficits; participation
MeSH Terms: conditions — Neuromuscular Diseases; Cerebral Palsy; Down Syndrome; Autistic Disorder; Motor Skills Disorders | interventions — Equine-Assisted Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment group (Experimental): Children between 5-17 years who have balance deficits related to any movement disorder (preferably neuromuscular)
  Interventions: Other: Hippotherapy

INTERVENTIONS:
Other: Hippotherapy — Children will receive treatment by a licensed physical therapist using hippotherapy as the treatment strategy. This includes sitting on a horse who's movement is controlled by a horse leader, with the PT directing the movements required of the horse, as well as supplying supplemental cues to the participant. Alternative positions (such as sitting backward and sideways) may also be used during the treatment session.

SUMMARY:
The purpose of this study is to determine if adding hippotherapy treatment will improve balance for children ages 5-17 who have disabilities such as cerebral palsy and down syndrome. We also want to find out if by improving their balance the children increase their participation in age appropriate activities.

DETAILED DESCRIPTION:
The primary purpose of this study is to determine the effects of hippotherapy on the balance of children with developmental disorders that cause mild to moderate balance problems. The secondary purpose is to determine if the use of hippotherapy also improves perceived functional abilities and thus quality of life as measured by the pediatric balance scale and Activities Scale for Kids (respectively)

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 5 and 17
* have a neuromuscular diagnosis or confirmed difficulties with balance
* be able to stand 4 seconds without an assistive device
* be able to follow testing instructions
* must be under 250 pounds
* be able to attend a minimum 10/12 sessions.

Exclusion Criteria:

* any compounding orthopedic or medical condition not related to the primary developmental diagnosis.
* previous hippotherapy intervention or therapeutic riding experience
* allergies or aversion to horses.
* refusal of parents to sign the therapeutic riding center's liability release form
* any new treatments (includes therapies, drugs, or other complementary treatments) within one month of the start of the study or plans for new treatments during the intervention period
* lack of a physician referral for physical therapy

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2006-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Pediatric Balance Scale | 8-9 weeks
  The Pediatric Balance Scale (PBS) is a standardized 14 item test of various component activities related to balance. It is a modified child version of the adult Berg Balance Scale. The PBS has high total score test-retest reliability of ICC (3,1) =0.998, as well as good interrater reliability (ICC(3,1) = 0.997).1

SECONDARY OUTCOMES:
Activities Scale for Kids | 8-9 weeks
  Activities Scale for Kids - Participation (ASKp) is a self-administered 30 item questionaire that measures the impact of children's disability to overall function and participation within relevant environments. It correlates well with parent reports on the Childhood Health Assessment Questionnaire (r=0.81, p<0.000) and clinician observations of children's function (ICC=0.92, p<0.000).

CONTACTS AND LOCATIONS:
Overall Officials: Debbie J Silkwood-Sherer, PT, DHS, Principal Investigator — Central Michigan University
Locations (1):
- CHUM Therapeutic Riding Center, Dansville, Michigan, United States

REFERENCES:
- [Background] McGibbon NH, Benda W, Duncan BR, Silkwood-Sherer D. Immediate and long-term effects of hippotherapy on symmetry of adductor muscle activity and functional ability in children with spastic cerebral palsy. Arch Phys Med Rehabil. 2009 Jun;90(6):966-74. doi: 10.1016/j.apmr.2009.01.011. PMID 19480872
- [Background] Casady RL, Nichols-Larsen DS. The effect of hippotherapy on ten children with cerebral palsy. Pediatr Phys Ther. 2004 Fall;16(3):165-72. doi: 10.1097/01.PEP.0000136003.15233.0C. PMID 17057544
- [Background] Benda W, McGibbon NH, Grant KL. Improvements in muscle symmetry in children with cerebral palsy after equine-assisted therapy (hippotherapy). J Altern Complement Med. 2003 Dec;9(6):817-25. doi: 10.1089/107555303771952163. PMID 14736353
- [Background] Silkwood-Sherer D, Warmbier H. Effects of hippotherapy on postural stability, in persons with multiple sclerosis: a pilot study. J Neurol Phys Ther. 2007 Jun;31(2):77-84. doi: 10.1097/NPT.0b013e31806769f7. PMID 17558361
- [Result] Silkwood-Sherer D. Hippotherapy as an Intervention to Improve Postural Control of Children with Movement Disorders. Dev Med Child Neurol 51(S5):18-19, 2009 [abstract]
- [Derived] Silkwood-Sherer DJ, Killian CB, Long TM, Martin KS. Hippotherapy--an intervention to habilitate balance deficits in children with movement disorders: a clinical trial. Phys Ther. 2012 May;92(5):707-17. doi: 10.2522/ptj.20110081. Epub 2012 Jan 12. PMID 22247403
- See also: Non profit organization that provides education, standards, terminology for physical, occupational and speech language pathologists using hippotherapy as part of their practice. — http://www.americanhippotherapyassociation.org